CLINICAL TRIAL: NCT04796766
Title: Establishment of a Human Electrophysiological Model to Quantify the Calcitonin Gene-related Peptide (CGRP)-Related Axon Reflex of Trigeminal Afferents and Its Evaluation as a Clinical Tool to Assess and Predict Treatment Effects of Migraine Prophylaxis
Brief Title: Human Electrophysiological Model to Quantify the CGRP-related Axon Reflex of Trigeminal Afferents
Acronym: MiPro-CGRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: MiPro-CGRP
Record Dates: First submitted 2021-03-01; First posted 2021-03-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Migraine
Keywords: Migraine; Calcitonin gene-related peptide (CGRP); Evoked flare response
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Experimental): HFS / LFS in healthy volunteers at two different points in time
  Interventions: Diagnostic Test: High frequency stimulation (HFS); Diagnostic Test: Low-frequency sinusoidal transcutaneous stimulation (sLFS)
- Migraine patients (Experimental): HFS / LFS in migraine patients at a single point in time
  Interventions: Diagnostic Test: High frequency stimulation (HFS); Diagnostic Test: Low-frequency sinusoidal transcutaneous stimulation (sLFS)
- Patients with Botulinum toxin or CGRP-targeted therapy (Experimental): HFS / LFS before and under treatment with Botulinum toxin or CGRP-targeted therapy
  Interventions: Diagnostic Test: High frequency stimulation (HFS); Diagnostic Test: Low-frequency sinusoidal transcutaneous stimulation (sLFS)

INTERVENTIONS:
Diagnostic Test: High frequency stimulation (HFS) — Electrical stimuli via circular electrode array. The electrode array serves as cathode placed above the eyebrow. A surface electrode (anode) will be placed on the temple. Electrical stimuli will be applied via a constant current stimulator. The stimulus intensity for the electrophysiological protocol is adjusted to the 10-fold of the detection threshold. A number of 5 electrical pulses (2 ms, 100 Hertz (Hz)), 10 second intervals.
Diagnostic Test: Low-frequency sinusoidal transcutaneous stimulation (sLFS) — Stimulation of C-nociceptors with constant current stimulator. Electrodes (placed on the proband's forehead. Stimulation by sine wave pulses of 250 ms duration (4 Hz), intensities inducing a pain intensity of 50/100 on a visual analogue scale from 0-100.

SUMMARY:
The proposed project aims at establishing Calcitonin gene-related peptide (CGRP)-Related Axon Reflex of Trigeminal Afferents as a neurophysiological biomarker for migraine.

DETAILED DESCRIPTION:
The proposed project aims at establishing a neurophysiological biomarker for migraine. Migraine is one of the world's most disabling diseases and its prophylactic treatment is time and cost-consuming. Since each patient responds differently and unpredictably to preventive medication, physicians are forced to try prophylactic drugs one by one. Recently, a new group of therapeutic agents targeting the neuropeptide Calcitonin gene-related peptide (CGRP) has been launched for migraine treatment. CGRP is stored in trigeminal afferents and released to meningeal blood vessels during acute migraine attacks leading to a vasodilating response. In an experimental setting, the release of CGRP from afferent nerve fibers in the skin can be induced by transdermal electrical stimulation. The subsequently evoked skin erythema, called 'flare reaction', can be quantified by laser Doppler imaging techniques. Never before, research studies used this experimental model in either trigeminally innervated skin or migraine patients. I therefore propose to establish this model to 1) test the specificity of an evoked 'flare response' in the trigeminal territory for the pathophysiology of migraine, 2) investigate the effect of CGRP-targeting anti-migraine drugs on this outcome parameter and 3) evaluate the impact of this model to predict the treatment response to drugs interfering with the CGRP-pathway. This study is a highly innovative approach towards tailored migraine treatment.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers (Study Arm 1 and 2):

* age ≥ 18 years
* good German language skills
* no history of head trauma
* no history of neurologic disease
* no primary headache disorder (e.g. migraine, episodic or chronic tension type headache, cluster headache)
* no regular drug intake (except for oral contraceptives)

Migraine patients need to match the following criteria (Study Arm 2 and 3):

* age ≥ 18 years
* good German language skills
* fulfilling the diagnostic criteria for either episodic or chronic migraine with or without aura according to the international classification of headache disorders (ICHD) 3rd edition
* history of migraine > 1 year
* keeping a headache diary for a minimum of 3 months prior to the study

Exclusion Criteria:

Healthy volunteers and migraine patients under the following conditions will be excluded:

* Chronic pain syndromes (e.g. low back pain, osteoarthritis, painful neuropathy, rheumatoid arthritis)
* Acute pain (e.g. pain due to acute skin injury, menstrual pain, acute toothache). In this case, a measurement can only be performed after complete remission of pain and at least 48 hours after intake of acute pain medication (e.g. triptans, non-steroidal anti-inflammatory drug (NSAID)).
* history of treatment with agents targeting the CGRP pathway (e.g. erenumab) < 3 months before the study
* history of treatment with Botulinum toxin < 9 months before the study
* Diseases of the skin involving the skin at face and forehead
* Pregnancy or breast feeding
* Subjects lacking capacity for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intensity of axonal flare reaction | Day 1
  Axon reflex erythema of stimulated C-nociceptors measured in Flux (luminous flux) values 0 - 100.

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid Schuh-Hofer, Prof. Dr., Principal Investigator — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No